CLINICAL TRIAL: NCT03606499
Title: Effectiveness of Ustekinumab in Patients Suffering From Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis) With Extra-intestinal Manifestations or Immune-mediated Inflammatory Diseases in a Real-world Setting
Brief Title: Real-world Effectiveness of Ustekinumab in Participants Suffering From Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis) With Extra-intestinal Manifestations or Immune-mediated Inflammatory Diseases
Acronym: TENOR
Status: Completed | Type: Observational
Sponsor: Janssen Cilag S.A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108498; CNTO1275CRD4012 (Other: Janssen Cilag S.A.S., France)
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease (IBD) Participants with EIMs and/or IMIDs: IBD (Crohn's Disease [CD] or Ulcerative Colitis [UC]) participants with suspected extra-intestinal manifestations (EIMs) and/or one or more immune-mediated inflammatory diseases (IMIDs) will be enrolled into the study to assess effectiveness of ustekinumab on EIMs and/or IMIDs associated with IBD (both CD and UC). Participants will receive ustekinumab at study entry (Week 0) as treatment for IBD according to standard clinical practice and will be followed up to 24 weeks (+/- 3 weeks). Only data available per clinical practice will be collected within this study.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — No study treatment will be administered as a part of this study. Participants who are initiating the treatment with ustekinumab, will be observed according to standard clinical practice.

SUMMARY:
The purpose of this study is to assess the effectiveness of ustekinumab on extra-intestinal manifestations (EIMs) and immune-mediated inflammatory diseases (IMIDs) associated with inflammatory bowel disease (IBD) (both Crohn's Disease [CD] and Ulcerative Colitis [UC]).

ELIGIBILITY:
Inclusion Criteria:

* With a confirmed diagnosis of CD or UC
* With at least one EIM of interest (cutaneous: pyoderma gangrenosum; erythema nodosum, articular: axial spondyloarthritis and peripheral spondyloarthritis with and without psoriasis, dactylitis, enthesitis; ocular: uveitis) and/or at least one IMIDs of interest (cutaneous: psoriasis, atopic dermatitis, hidradenitis suppurativa), suspected or confirmed, that is active at the time of screening
* Starting ustekinumab as a biologic therapy for CD or UC treatment independently of their enrollment into the study
* Using ustekinumab according to the SmPC
* Only for participants with CD: has had an inadequate response with or lost response to or be intolerant to conventional therapy including azathioprine, 6-mercaptopurine or corticosteroids or; at least one tumor necrosis factor (TNF) blocker (adalimumab, infliximab). Only for participants with UC: Have had an inadequate response with, lost response to, or were intolerant to either conventional including azathioprine, 6-mercaptopurine or corticosteroids or a biologic

Exclusion Criteria:

* Participants suffering from a psoriasis induced by a biological therapy at inclusion (including TNF blocker) or participant presenting an active psoriasis that was diagnosed before the time of inflammatory bowel disease (IBD) diagnosis
* Participants currently enrolled in an investigational study (or have been in the past 2 months) or are unwilling or not able to understand or provide their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be participants with a confirmed diagnosis of moderate to severe Crohn's Disease (CD) or Ulcerative Colitis (UC) with at least one extra-intestinal manifestation (EIM) or immune-mediated inflammatory disease (IMID) of interest and for which a treatment with ustekinumab is indicated according to the clinical practice and Summary of Product Characteristics (SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Clinical Response (CR) on at Least one Extra-intestinal Manifestation/Immune-mediated Inflammatory Disease (EIM/IMID) Associated with Inflammatory Bowel Disease (IBD) at Week 24 | Week 24
  CR will be determined based on the measures collected by the investigators which will be assessed by the specialists based on these parameters: 2 points reduction in physician global assessment (PGA) score or PGA 0 or 1 (0= clear to 5=very severe) achieved for cutaneous disease, or resolution of lesions for Erythema nodosum (dermatology); decrease of 50 percent (%) of ankylosing spondylitis disease activity index (BASDAI) (1=no problem to 10=worst problem) for axial spondyloarthritis (SpA); disease activity score (DAS)28 (derived from 4 items with score <2.6 [disease remission] and >5.1 [severe disease activity]) of moderate and good response achieved in peripheral SpA plus 2 points reduction in PGA score or PGA 0 or 1 achieved in case of associated psoriasis; resolution of dactylitis, decrease of 50% of Leeds enthesitis index [LEI-6] score which ranges from 0 [pain/tenderness absent] to1 [pain/tenderness present] for enthesitis, (rheumatology); resolution of uveitis (ophthalmology).

SECONDARY OUTCOMES:
Percentage of Participants with Change from Baseline in Clinical Response for Crohn's Disease (CD) as Measured by Harvey-Bradshaw Index (HBI) | Baseline, Week 16 and Week 24
  HBI is defined as total HBI score of 4 points or less. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well-being.
Percentage of Participants Achieving Remission for CD as Measured by HBI | Up to Week 24
  Percentage of participants achieving remission for CD will be measured using the HBI Score less than or equal to (<= 4). HBI remission is defined as total HBI score of 4 points or less. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well-being.
Change from Baseline in Partial Mayo Score | Baseline, Week 16 and Week 24
  Mayo scoring system is used for assessment of ulcerative colitis activity. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, physician's global assessment, and endoscopy findings) each ranging from 0 to 3. Partial Mayo score is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, and physician's global assessment) and ranges from 0 to 9 points. Higher score indicates severe disease. Change from baseline in the Partial Mayo Score of at least 3 points and at least 30 percent, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1 will be reported.
Percentage of Participants Achieving Remission for UC as Measured by Partial Mayo Score (Score of <=2) | Up to Week 24
  Percentage of participants achieving remission for UC will be measured using the Partial Mayo score Score less than or equal to <=2). Partial Mayo score is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, and physician's global assessment) and ranges from 0 to 9 points. Higher score indicates severe disease.
Change from Baseline in the Presence of Extra Intestinal Manifestations (EIMS) or Immune-Mediated Inflammatory Diseases (IMIDs) | Baseline and Week 24
  Change from baseline in the presence of Extra Intestinal Manifestations (EIMs)/ Immune-Mediated Inflammatory Diseases (IMIDs) for its severity/activity will be determined.
Work Productivity and Activity Impairment (WPAI) Questionnaire | Baseline, Weeks 16 and Week 24
  The WPAI is a validated, self-administered questionnaire that assesses work and activity impairment during the past 7 days due to IBD. The WPAI score ranges from 0 to10. Score 0 means IBD had no effect on work and score 10 indicates because of IBD, could not work at all.
Short Inflammatory Bowel Disease Questionnaire Score (Short IBDQ) | Baseline, Weeks 16 and 24
  Short IBDQ is a health-related quality of life tool (HRQoL) to assess quality of life in adult participants with inflammatory bowel disease (IBD) having only 10 items with 4 domains: digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbance (3 items), and social function (2 items). Participants are asked to recall symptoms and quality of life from the last 2 weeks and rate each item on a 7-point Likert scale (1=all of the time; 2=most of the time; 3=a good bit of the time; 4=some of the time; 5=a little bit of the time; 6=hardly any of the time; 7=none of the time). Total score is calculated by adding the scores from each domain; the total score ranges from 10 to 70, where minimum score =10 (poor HRQoL) and maximum score =70 (good HRQoL).
Functional Assessment of Chronic Illness Therapy Scale (FACIT) | Baseline, Weeks 16 and 24
  FACIT-F scale is a 13 item fatigue scale with a 7 day recall period. It measures the level of fatigue during the usual daily activities. The level of fatigue is measured on a 4 point Likert scale (0=very much fatigued to 4=not at all fatigued). Total FACIT score is the sum of 13 items, ranging from 0 (not at all) to 52 (very much). Higher scores represent better outcomes.
Inflammatory Bowel Disease-Disability Index (IBD-DI) | Baseline, Weeks 16 and 24
  The IBD-DI consists of 28 items that evaluate the 5 domains of overall health, body function, body structures, activity participation and environmental factors. Each item response is graded from 0 to 4 for each area evaluated (0 = very good; 1 = Good; 2 = medium; 3 = Bad; 4 = Very bad). The final composite score representative of the overall degree of disability ranging from -80 (maximum degree of disability) to 22 (no disability).
Number of Participants with Adverse Events | Up to 37 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of IBD Related Medical Visits | Week 24
  Number of IBD related medical visits as a part of medical resources utilization will be reported.
Number of Days of IBD Related Hospitalization with Surgery | Week 24
  Number of days of IBD related hospitalization with surgery (defined as number of days from the day of admission to discharge) as a part of medical resources utilization will be reported.
Number of Days of IBD Related Hospitalization Without Surgery | Week 24
  Number of days of IBD related hospitalization without surgery (defined as number of days from the day of admission to discharge) as a part of medical resources utilization will be reported.
Number of IBD Related Emergency Visits | Week 24
  Number of IBD related emergency visits as a part of medical resources utilization will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag S.A.S., France Clinical Trial, Study Director — Janssen Cilag S.A.S.
Locations (1):
- CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy, France